CLINICAL TRIAL: NCT05419726
Title: Brown Adipose Tissue Activity in Response to Semaglutide Administered to Obese Subjects.
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Preethi Srikanthan, MD, MS, Professor, University of California, Los Angeles
Other Study IDs: 22-000718
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Semaglutide Injectable Product (not provided by the study) — Study Procedure:
  Subjects that are to be started on semaglutide by their physician will be invited to participate in the study. If the subject is eligible and signs the consent form they will be enrolled in the study. There are three (3) study visits including Baseline/Visit 1 (prior to starting semaglutide), Visit 2 (at week 2-4) and Visit 3 (at week 18-20). The subjects undergo these tests at each visit: weight circumference measured, BMR testing, thermal imaging of BAT, and perform a 24 hour food recall.

SUMMARY:
Glucagon like peptide (GLP-1) agonists, such as liraglutide, exenatide, and semaglutide, have been increasingly used as a medication to address the current twin epidemics of diabetes and obesity. Their activities include increasing insulin production by pancreatic beta cells, improving insulin sensitivity in muscles and weight loss. The mechanisms underpinning the weight loss caused by GLP-1 agonists have not yet been fully elucidated, but brown adipose tissue (BAT) appears to play an important role.

We propose to assess BAT activity, using infrared thermography camera images, before individuals start weekly administration of semaglutide, at week 2-4, and week 18-20. We hypothesize that this GLP-1 agonist, semaglutide, will cause an increase in BAT activity and a corresponding increase in basal metabolic rate.

DETAILED DESCRIPTION:
Background and Rationale:

Glucagon like peptide (GLP-1) agonists, such as liraglutide, exenatide, and semaglutide, have been increasingly used as a medication to address the current twin epidemics of diabetes and obesity. Their activities include increasing insulin production by pancreatic beta cells, improving insulin sensitivity in muscles and weight loss. The mechanisms underpinning the weight loss caused by GLP-1 agonists have not yet been fully elucidated, but brown adipose tissue (BAT) appears to play an important role.

BAT is a type of adipose tissue which predominates in infants to allow thermoregulation through adaptive thermogenesis, but it is also present in adults. BAT activity also increases insulin sensitivity and whole body energy expenditure, and thus has the potential to treat type 2 diabetes and obesity. Bilateral supraclavicular and axillary BAT account for approximately two thirds of total body BAT content. Although the precise role of BAT in human metabolism and energy balance is unknown, a clear link exists between obesity and BAT dysfunction in humans.

It has been hypothesized that the prominent weight loss activity of GLP-1 agonists in humans is the result of BAT activation. However, studies with various GLP-1 agonists have been equivocal.

With more powerful GLP-1 agonists such as semaglutide entering in clinical practice, a better understanding of the relationship between GLP-1 and BAT is important. If BAT activity is found to be clinically significant as a mechanism of action of GLP-1 agonists, then the addition of adjuvants which enhance BAT activity could optimize the benefit of these medications.

Currently, the main methods available to assess BAT activity are PET-CT with 18F-fluorodeoxyglucose, single-photon-emission CT scanning with tracers such as 123 I-meta-iodobenzylguanidine or 99mTc-tetrofosmin, and/or tissue biopsy 17-19.These techniques have distinct disadvantages as they are expensive and require either the administration of radiopharmaceuticals or tissue sampling. Their utility is, therefore, greatly limited as they can only be conducted on a very small number of subjects and are unable to provide indices of BAT function in real-time. Symonds et al demonstrated the feasibility of using infrared thermography as a safe, reproducible, and robust technique for measuring the temperature of the skin overlying BAT depots in the supraclavicular region and quantifying BAT thermogenesis induced by a cold challenge.

We propose to assess BAT activity, using infrared thermography camera images, before individuals start weekly administration of semaglutide, at week 2- 4, and week 18-20. We hypothesize that this GLP-1 agonist, semaglutide, will cause an increase in BAT activity and a corresponsing increase in basal metabolic rate.

Utilizing a reproducible and non invasive measure of BAT activity, we hope to gain better understanding of BAT activity in concert with the metabolic status of patients commenced on semaglutide. This will not only allow insights into the mechanism of achieving weight loss with semaglutide, it will also allow better understanding of the importance of BAT activity manipulation in the therapy for obesity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled to start semaglutide for weight loss (drug not provided by or paid for by the study)
* >18 years of age and willing to participate
* Male or post-menopausal females

Exclusion Criteria:

* History of prior neck surgery and /or neck irradiation

  * Use of beta blocker agents
  * Use of any other glucose lowering medication
  * History of neuropathic disorders (e.g. diabetic neuropathy)
  * Diabetic patients
  * Individuals without normal thyroid function
  * Individuals with cancer
  * Any significant chronic disease or renal, hepatic or endocrine disease
  * Current smokers
  * Inability of patient to provide consent either for medical reasons or psychiatric reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult >18 years of age, non-diabetic but obese The study is a non-randomized single center study. Subjects who are to be started by their physician or endocrinologist on semaglutide for weight loss, and are willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
change in supraclavicular temperature with cold exposure | 20weeks
  delta temperature
change in caloric intake | 20weeks
  caloric intake
basal metabolic rate | 20 weeks
  basal metabolic rate (ml O2/min or joule per hour per kg body mass)

CONTACTS AND LOCATIONS:
Overall Officials: Preethi Srikanthan, MD, Principal Investigator — Principal Investigator
Locations (1):
- UCLA Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Garcia I, Milbank E, Dieguez C, Lopez M, Contreras C. Glucagon, GLP-1 and Thermogenesis. Int J Mol Sci. 2019 Jul 13;20(14):3445. doi: 10.3390/ijms20143445. PMID 31337027
- [Background] Stafeev I, Sorkina E, Koksharova E, Tumanyan T, Sklyanik I, Menshikov M, Mayorov A, Parfyonova Y, Shestakova M. The Effects of Glucagon-Like Peptide Type 1 (GLP-1) and its Analogues in Adipose Tissue: Is there a way to Thermogenesis? Curr Mol Med. 2021;21(7):527-538. doi: 10.2174/1566524020666201201095029. PMID 33261539
- [Background] Cypess AM, Lehman S, Williams G, Tal I, Rodman D, Goldfine AB, Kuo FC, Palmer EL, Tseng YH, Doria A, Kolodny GM, Kahn CR. Identification and importance of brown adipose tissue in adult humans. N Engl J Med. 2009 Apr 9;360(15):1509-17. doi: 10.1056/NEJMoa0810780. PMID 19357406
- [Background] Blondin DP, Labbe SM, Noll C, Kunach M, Phoenix S, Guerin B, Turcotte EE, Haman F, Richard D, Carpentier AC. Selective Impairment of Glucose but Not Fatty Acid or Oxidative Metabolism in Brown Adipose Tissue of Subjects With Type 2 Diabetes. Diabetes. 2015 Jul;64(7):2388-97. doi: 10.2337/db14-1651. Epub 2015 Feb 12. PMID 25677914
- [Background] Lee P, Smith S, Linderman J, Courville AB, Brychta RJ, Dieckmann W, Werner CD, Chen KY, Celi FS. Temperature-acclimated brown adipose tissue modulates insulin sensitivity in humans. Diabetes. 2014 Nov;63(11):3686-98. doi: 10.2337/db14-0513. Epub 2014 Jun 22. PMID 24954193
- [Background] Ong FJ, Ahmed BA, Oreskovich SM, Blondin DP, Haq T, Konyer NB, Noseworthy MD, Haman F, Carpentier AC, Morrison KM, Steinberg GR. Recent advances in the detection of brown adipose tissue in adult humans: a review. Clin Sci (Lond). 2018 May 25;132(10):1039-1054. doi: 10.1042/CS20170276. Print 2018 May 31. PMID 29802209
- [Background] Beiroa D, Imbernon M, Gallego R, Senra A, Herranz D, Villarroya F, Serrano M, Ferno J, Salvador J, Escalada J, Dieguez C, Lopez M, Fruhbeck G, Nogueiras R. GLP-1 agonism stimulates brown adipose tissue thermogenesis and browning through hypothalamic AMPK. Diabetes. 2014 Oct;63(10):3346-58. doi: 10.2337/db14-0302. Epub 2014 Jun 10. PMID 24917578
- [Background] Lee SJ, Sanchez-Watts G, Krieger JP, Pignalosa A, Norell PN, Cortella A, Pettersen KG, Vrdoljak D, Hayes MR, Kanoski SE, Langhans W, Watts AG. Loss of dorsomedial hypothalamic GLP-1 signaling reduces BAT thermogenesis and increases adiposity. Mol Metab. 2018 May;11:33-46. doi: 10.1016/j.molmet.2018.03.008. Epub 2018 Mar 21. PMID 29650350
- [Background] Lockie SH, Heppner KM, Chaudhary N, Chabenne JR, Morgan DA, Veyrat-Durebex C, Ananthakrishnan G, Rohner-Jeanrenaud F, Drucker DJ, DiMarchi R, Rahmouni K, Oldfield BJ, Tschop MH, Perez-Tilve D. Direct control of brown adipose tissue thermogenesis by central nervous system glucagon-like peptide-1 receptor signaling. Diabetes. 2012 Nov;61(11):2753-62. doi: 10.2337/db11-1556. Epub 2012 Aug 28. PMID 22933116
- [Background] Oliveira FCB, Bauer EJ, Ribeiro CM, Pereira SA, Beserra BTS, Wajner SM, Maia AL, Neves FAR, Coelho MS, Amato AA. Liraglutide Activates Type 2 Deiodinase and Enhances beta3-Adrenergic-Induced Thermogenesis in Mouse Adipose Tissue. Front Endocrinol (Lausanne). 2022 Jan 4;12:803363. doi: 10.3389/fendo.2021.803363. eCollection 2021. PMID 35069450
- [Background] Krieger JP, Santos da Conceicao EP, Sanchez-Watts G, Arnold M, Pettersen KG, Mohammed M, Modica S, Lossel P, Morrison SF, Madden CJ, Watts AG, Langhans W, Lee SJ. Glucagon-like peptide-1 regulates brown adipose tissue thermogenesis via the gut-brain axis in rats. Am J Physiol Regul Integr Comp Physiol. 2018 Oct 1;315(4):R708-R720. doi: 10.1152/ajpregu.00068.2018. Epub 2018 May 30. PMID 29847161
- [Background] Harder H, Nielsen L, Tu DT, Astrup A. The effect of liraglutide, a long-acting glucagon-like peptide 1 derivative, on glycemic control, body composition, and 24-h energy expenditure in patients with type 2 diabetes. Diabetes Care. 2004 Aug;27(8):1915-21. doi: 10.2337/diacare.27.8.1915. PMID 15277417
- [Background] van Eyk HJ, Paiman EHM, Bizino MB, IJzermans SL, Kleiburg F, Boers TGW, Rappel EJ, Burakiewicz J, Kan HE, Smit JWA, Lamb HJ, Jazet IM, Rensen PCN. Liraglutide decreases energy expenditure and does not affect the fat fraction of supraclavicular brown adipose tissue in patients with type 2 diabetes. Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):616-624. doi: 10.1016/j.numecd.2019.12.005. Epub 2019 Dec 13. PMID 32127340
- [Background] Horowitz M, Flint A, Jones KL, Hindsberger C, Rasmussen MF, Kapitza C, Doran S, Jax T, Zdravkovic M, Chapman IM. Effect of the once-daily human GLP-1 analogue liraglutide on appetite, energy intake, energy expenditure and gastric emptying in type 2 diabetes. Diabetes Res Clin Pract. 2012 Aug;97(2):258-66. doi: 10.1016/j.diabres.2012.02.016. Epub 2012 Mar 24. PMID 22446097
- [Background] Bradley DP, Kulstad R, Racine N, Shenker Y, Meredith M, Schoeller DA. Alterations in energy balance following exenatide administration. Appl Physiol Nutr Metab. 2012 Oct;37(5):893-9. doi: 10.1139/h2012-068. Epub 2012 Jun 26. PMID 22735035
- [Background] Janssen LGM, Nahon KJ, Bracke KFM, van den Broek D, Smit R, Sardjoe Mishre ASD, Koorneef LL, Martinez-Tellez B, Burakiewicz J, Kan HE, van Velden FHP, Pereira Arias-Bouda LM, de Geus-Oei LF, Berbee JFP, Jazet IM, Boon MR, Rensen PCN. Twelve weeks of exenatide treatment increases [18F]fluorodeoxyglucose uptake by brown adipose tissue without affecting oxidative resting energy expenditure in nondiabetic males. Metabolism. 2020 May;106:154167. doi: 10.1016/j.metabol.2020.154167. Epub 2020 Jan 23. PMID 31982480
- [Background] Fukuchi K, Ono Y, Nakahata Y, Okada Y, Hayashida K, Ishida Y. Visualization of interscapular brown adipose tissue using (99m)Tc-tetrofosmin in pediatric patients. J Nucl Med. 2003 Oct;44(10):1582-5. PMID 14530470
- [Background] Symonds ME, Henderson K, Elvidge L, Bosman C, Sharkey D, Perkins AC, Budge H. Thermal imaging to assess age-related changes of skin temperature within the supraclavicular region co-locating with brown adipose tissue in healthy children. J Pediatr. 2012 Nov;161(5):892-8. doi: 10.1016/j.jpeds.2012.04.056. Epub 2012 Jun 5. PMID 22677567
- [Background] Thackeray JT, Beanlands RS, Dasilva JN. Presence of specific 11C-meta-Hydroxyephedrine retention in heart, lung, pancreas, and brown adipose tissue. J Nucl Med. 2007 Oct;48(10):1733-40. doi: 10.2967/jnumed.107.043570. Epub 2007 Sep 14. PMID 17873125
- [Background] Robinson L, Ojha S, Symonds ME, Budge H. Body mass index as a determinant of brown adipose tissue function in healthy children. J Pediatr. 2014 Feb;164(2):318-22.e1. doi: 10.1016/j.jpeds.2013.10.005. Epub 2013 Nov 14. PMID 24238856